CLINICAL TRIAL: NCT05548686
Title: Benefits of Adapted Physical Activity for Chronic Osteoarticular Pain in Patients With Multiple Myeloma
Acronym: ALGOMYELOMOV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-163; 2020-A02599-30 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2021-12-07; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2021-12

CONDITIONS: Multiple Myeloma; Adapted Physical Activity; Chronic Pain
MeSH Terms: conditions — Multiple Myeloma; Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted Physical Activity (Experimental): Patients benefiting from adapted physical activity
  Interventions: Other: adapted physical activity

INTERVENTIONS:
Other: adapted physical activity — 3 sessions of adapted physical activity per week during 12 weeks for each patient

SUMMARY:
Pain is one of the most frequent symptoms leading patients to consult a doctor, particularly in rheumatology and cancerology. When it becomes chronic, pain is the cause of a major emotional and physical invasion, with harmful repercussions on the family, social and professional levels. It is therefore necessary to be able to propose different therapies.

For many years, non-medicinal techniques have been proving their benefits and their central role in the treatment of chronic pain. Physical activity has been widely demonstrated in the literature to have considerable physical benefits (reduced risk of hypertension, vascular accidents, diabetes, improved bone condition, weight control, etc.) but also psychological benefits. However, according to the WHO, nearly 31% of adults aged 15 and over were not physically active in 2008. Physical inactivity is considered the 4th leading risk factor for death in the world. It is estimated to be the main cause of 21 to 25% of breast and colon cancers.

The investigators therefore propose a feasibility study, interventional, with minimal risks and constraints, evaluating the effectiveness of adapted physical activity in chronic pain related to a pathology little studied in this field of management: multiple myeloma. This study will include about 15 patients with residual pain 3 months after the end of their induction chemotherapy treatment.

Adapted Physical Activity sessions will be performed for 12 weeks. The evaluation of the expected benefits on pain and its consequences (cognitive, emotional, behavioral, physical ...) will be done through simple and validated questionnaires as well as on the evolution of the consumption of analgesics. The expected duration of the study will be one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain related to multiple myeloma, which has been evolving for more than 3 months and whose intensity is assessed with a VAS > 30/100

  * Patients who have completed more than 3 months of induction chemotherapy for Multiple Myeloma.
  * Patients not eligible for bone marrow transplantation.
  * Patient able to read, understand French and self-assess their pain on the VAS
  * Patient followed in the haematology department of the Caen University Hospital and living in Calvados

Exclusion Criteria:

* Patients with absolute contraindications to Adapted Physical Activity.

  * Unstable angina
  * Decompensated heart failure
  * Complex ventricular rhythm disorders
  * Severe uncontrolled hypertension
  * PAH > 60mmHg
  * Presence of large or pedunculated intra-cavity thrombus
  * Acute pericardial effusion
  * Severe obstructive cardiomyopathy
  * Tight and/or symptomatic aortic stenosis
  * Recent thrombophlebitis with or without pulmonary embolism
  * Diabetes with plantar perforating disease for activities involving the lower limbs
* Patient eligible for a bone marrow transplant.
* Patients with a major and/or potentially dangerous osteolytic lesion.
* Patients who do not meet the criteria for "moderate" functional impairment (assessed at the inclusion visit). defined by the HAS in 2019
* Pregnant or lactating woman.
* Minor patient.
* Patient under legal protection.
* Patient who does not read or understand French.
* Patient undergoing physiotherapy at the time of inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of adapted physical activity on the intensity of chronic pain related to multiple myeloma | difference between Month 0, Month 3, Month 6
  Evaluation of the pain intensity with the visual analogue scale from 0 to 100 (with the help of the ruler) over time

SECONDARY OUTCOMES:
Evaluate the impact of adapted physical activity on pain | difference between Month 0, Month 3, Month 6
  Brief Pain Inventory (BPI), 7 items from 0 (no discomfort) to 10 (complete discomfort) on the impact of the pain (sleep, enjoyment of life, relationships with others, work, general activity, ability to walk, mood. Score for each item.
To evaluate the impact of APA on the consumption of analgesics. | difference between Month 0, Month 3, Month 6
  Percentage of patients who reduced their treatment at the end of follow-up
Evaluate the impact of adapted physical activity on catastrophizing | difference between Month 0, Month 3, Month 6
  Pain Catastrophization Scale (PCS) Questionnaires reporting the patient's thoughts when in pain (e.g., "I'm afraid to die") ranging from "not at all = 0" to "all the time = 4". Total score out of 52.
Evaluate the impact of adapted physical activity on anxiety and depression | difference between Month 0, Month 3, Month 6
  Assessment of anxiety and depression with the Hospital Anxiety and Depression Scale (HAD score) 14 items from 0 to 3: a total score from 0 to 42 and 2 other scores differentiating anxiety and depression
Evaluate the impact of adapted physical activity on sleep | difference between Month 0, Month 3, Month 6
  Sleep assessment wit the PSQI (Pittsburgh Sleep Quality Index) 19 self-report questions and 5 questions asked of the spouse or roommate (if any). Only the self-report questions are included in the score. The 19 self-report questions combine to give 7 "components" of the overall score, with each component receiving a score from 0 to 3. In all cases, a score of 0 indicates no difficulty while a score of 3 indicates severe difficulty. The 7 components of the score are added together to give an overall score ranging from 0 to 21 points, with 0 indicating no difficulty and 21 indicating major difficulty.
Evaluate the impact of adapted physical activity on physical activity | difference between Month 0, Month 3, Month 6
  Physical activity assessment with the International Physical Activity Questionnaire (IPAQ) 7 questions about daily physical activity in the last 7 days, distinguishing between time spent doing moderate-intensity physical activity (carrying light loads, vacuuming, cycling quietly, playing volleyball ...), high-intensity physical activity (carrying heavy loads, digging, mountain biking, playing soccer ...), and time spent walking and sitting. Depending on the intensity (converted into METs), duration and number of days in the week, a physical activity score is defined ranging from low, moderate to high.
Evaluate the impact of adapted physical activity on self-esteem | difference between Month 0, Month 3, Month 6
  Assessment of Self-esteem with Physical Self Inventory (ISP25) 25 items composed of 6 scales: at the general level, a global self-esteem scale with 5 items, of which 2 items are presented in positive form (items 1 and 2) and 3 items in negative form (items 7, 13 and 19); at the physical level, a perceived physical value scale with 5 positive items (2, 8, 14, 20 and 24) ; 4 other subscales correspond to the physical condition, evaluated on the basis of the endurance race with 5 items, of which 3 positive items (items 9, 15 and 21) and 2 negative items (items 3 and 25), the sports competence made up of 4 items in positive form (items 4, 10, 16, 22), the physical appearance made up of 3 items of which 1 positive item (item 11) and two negative items (items 5 and 17) and the strength with 3 positive items (items 6, 12 and 18). The scoring of the negative items is reversed.
Evaluate the impact of adapted physical activity on quality of life | difference between Month 0, Month 3, Month 6
  Assessment of quality of life with the Quality of Life Questionnaires in Cancer (QLQC30).
  28 questions with 4 items ranging from "not at all" to "a lot" and dealing with the evaluation of several parameters (current and during the past week): physical, social, cognitive, personal and psychological functioning, overall health status, fatigue, nausea vomiting, pain, dyspnea, insomnia, loss of appetite, constipation, diarrhea, ﬁncial problems. There are also 2 additional questions ranging from 1 "very poor" to 7 "excellent" on the overall quality of life felt by the patient. Measurement of the total quality of life score combining all 30 questions.